CLINICAL TRIAL: NCT04717193
Title: Laparoscopically Guided Rectus Sheath Block in Pediatric Appendicitis - a Randomized Control Trial
Brief Title: Laparoscopically Guided Rectus Sheath Block in Pediatric Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSB-001
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single-blind. Surgeon cannot be blinded to the intervention. Anesthesiologist, participants, parents, and nursing staff in the OR, recovery room, and ward will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectus Sheath Block (Experimental): Participants randomized to the experimental arm will receive a bilateral rectus sheath block which is additional to the standard of care (infiltration of 5mg (2mL) 0.25% bupivacaine with epinephrine around port site incisions). For rectus sheath block, use the formula Volume (ml) = 2mg/kg x weight (kg) divided by 2.5mg/ml - 6ml to a maximum of 14ml. Maximum total dose is 2mg/kg. Participants will be asked to rate their pain a total of 4 times for the study. Each occurrence is expected to take approximately 1-2 minutes to complete. There will be no additional follow-up required as part of the study. The 6 week follow-up visit is standard routine practice.
  Interventions: Drug: Rectus Sheath Block with 0.25% bupivicaine with 1:200 000 epinephrine
- Local Anesthetic (Active Comparator): Participants in the control arm will receive the standard care which is infiltration of 5mg (2mL) of 0.25% bupivacaine with epinephrine around port site incisions. Participants will be asked to rate their pain a total of 4 times for the study. Each occurrence is expected to take approximately 1-2 minutes to complete. There will be no additional follow-up required as part of the study. The 6 week follow-up visit is standard routine practice.
  Interventions: Procedure: Local Anesthetic Infiltration with 0.25% bupivicaine with 1:200 000 epinephrine

INTERVENTIONS:
Drug: Rectus Sheath Block with 0.25% bupivicaine with 1:200 000 epinephrine — Bilateral rectus sheath block plus infiltration local anesthetic at incision sites.
  Arms: Rectus Sheath Block
Procedure: Local Anesthetic Infiltration with 0.25% bupivicaine with 1:200 000 epinephrine — Infiltration of local anesthetic at incision sites.
  Arms: Local Anesthetic

SUMMARY:
The study will investigate the pain control effects of a rectus sheath block after laparoscopic surgery to remove the appendix. A rectus sheath block is the injection of local anesthetic (numbing agent) into the space between the muscles of the belly wall. Children having surgery for appendicitis age 8-17 at the Stollery Children's Hospital will be eligible to participate. Patients with complicated appendicitis (perforation or abscess), chronic pain, bleeding disorders, or inability to document pain scores will be excluded from this study.

Participants will be randomly assigned to either rectus sheath block or standard local anesthetic. The standard local anesthetic group will have local anesthetic (numbing agent) injected around their surgery cut sites. The rectus sheath block group will have this standard plus the rectus sheath block with local anesthetic. Participants, parents, anesthesiologists and nursing staff will not know which group the participant has been assigned to. The surgeon will know the group.

The same pain and nausea medications will be ordered for all participants after the surgery. Pain scores will be measured using the Faces Pain Scale - Revised tool. Participants will be asked to rate their pain in the recovery room, in their hospital room at 3 and 6 hours after the surgery and again before going home. This tool has been shown to be useful for rating children's pain levels. The study will also measure the amount of pain and nausea medications that participants are given during their surgery and recovery. Participants will see their surgeon at 6 weeks after their surgery where they will be asked about any problems after being discharged home. Data will be analyzed with a linear mixed model.

DETAILED DESCRIPTION:
Purpose:

To determine if a bilateral laparoscopically guided rectus sheath block improves pain control over conventional local anesthetic infiltration around port site incisions following laparoscopic appendectomy.

Hypothesis:

Bilateral rectus sheath block will improve post-operative pain scores following laparoscopic appendectomy for acute uncomplicated appendicitis.

Justification:

Children have significant pain after laparoscopic appendectomy and many receive post-operative opioids for analgesia. The Faces pain scale - revised (FPS-R) is a simple validated method of measuring post-operative pain in children. Ultrasound-guided bilateral rectus sheath block (RSB) has been shown to decrease pain scores in the early post-operative period following pediatric laparoscopic appendectomy and elective umbilical hernia repair.2,4 The use of image-guidance for needle placement has improved both achievement of appropriate anatomic location of the block as well as analgesia associated with the block. Under ultrasound guidance, this extra step requires additional equipment, time, and sometimes dedicated personnel to complete. The investigators propose a bilateral RSB performed intra-operatively under laparoscopic guidance may alleviate the need for these extra resources while achieving the desired analgesic effects.

The analgesic effect of the standard of care injection of local anesthesia is limited to the superficial layers of the abdominal wall. The rectus sheath block targets the nerves running within the fascia and provides a more complete block to the deep and superficial layers of the abdominal wall.

Objectives:

Primary Objective: Determine if intra-operative laparoscopic guided bilateral RSB improves self-reported post-operative pain scores at 3 hours post-operatively.

Secondary Objectives:

Determine if intra-operative laparoscopic guided bilateral RSB improves self-reported post-operative pain scores in the PACU, at 6 hours post-operatively, and prior to discharge home.

Determine if intra-operative bilateral laparoscopic guided bilateral RSB decreases intra-operative narcotic use, post-operative opioid use, and post-operative antiemetic use.

Research Methods/Procedures:

Randomization: Simple

Blinding: Single-blind. Surgeon cannot be blinded to the intervention. Anesthesiologist, participants, parents, and nursing staff in the OR, recovery room, and ward will be blinded.

Control: Standard of care infiltration of local anesthetic at incisions.

Treatment and standard care arms will run in parallel.

Standard Care: Intra-operative infiltration of 2ml of 0.25% Bupivacaine with 1:200 000 epinephrine at each port site incision.

Experimental Treatment: Bilateral RSB with up to 7ml of 0.25% Bupivacaine with 1:200 000 epinephrine plus 2ml infiltrated around each port site incision as in the standard care group. The total volume used will not exceed 20ml or 2mg/kg, whichever is lower.

Each participant will be followed in the recovery room and surgical ward and asked to report their pain level immediately after surgery, at 3 and 6 hours after surgery, and prior to discharge home. Each participant will have a scheduled follow up visit at 6 weeks with their operating surgeon where they will be asked about any complications experienced since discharge.

Participation will be voluntary. Participants will receive standard of care if they choose not to participate in the study. Informed consent will be obtained from the participant's parent or legal guardian by the operating surgeon or delegate pre-operatively. Participants will be asked to provide assent.

Plan for Data Analysis:

100 participants will be required with a target of 50 in each group. Sample size calculations were completed based on an estimated 20% effect size with consideration for a potential 10-15% dropout rate to achieve a power of 80% and alpha 5%. Effect size is estimated conservatively from data in previous studies showing an average 30% decrease in early post-operative pain scores.

Data will be analyzed in an intent to treat manner using a linear mixed model. We have undertaken an initial consultation with a WCHRI biostatistician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute uncomplicated appendicitis
* Age 8-17 years

Exclusion Criteria:

* Complicated appendicitis, perforation, abscess
* History of chronic pain condition or long-term analgesic use
* History of bleeding condition
* Condition preventing accurate documentation of post-operative pain scores using the FPS-R tool including severe developmental delay, psychiatric illness, or partially sighted or blindness
* Previous open abdominal surgery
* Presence of an abdominal prosthesis such as a gastrostomy tube or ventricular-peritoneal shunt device
* Allergy to bupivacaine or morphine

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Self-reported pain scores at 3 hours post-operatively | 3 hours
  Reported with Faces Pain Scale - Revised. Scale runs from 0-10 with 0 being no pain and 10 being the worst pain they have experienced.

SECONDARY OUTCOMES:
Self-reported pain scores in recovery room, at 6 hours post-operatively, and prior to discharge home | Immediately post-operatively to approximately 24 hours
  Reported with Faces Pain Scale - Revised. Scale runs from 0-10 with 0 being no pain and 10 being the worst pain they have experienced.
Intra-operative narcotic use in mg/kg morphine equivalents | Intra-operative
  Opioid medications administered intra-operatively
Post-operative narcotic use in mg/kg morphine equivalents | Approximately 24 hours
  Opioid medications administered post-operatively
Post-operative anti-emetic use mg/kg or ondansetron and dimenhydrinate | Approximately 24 hours
  Anti-emetic medications (ondansetron and dimenhydrinate) administered post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Troy Perry, MD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers. For inquiries relating to the study protocol or other supporting information, researchers are invited to contact the study's principal investigator.

REFERENCES:
- [Background] Dingeman RS, Barus LM, Chung HK, Clendenin DJ, Lee CS, Tracy S, Johnson VM, Dennett KV, Zurakowski D, Chen C. Ultrasonography-guided bilateral rectus sheath block vs local anesthetic infiltration after pediatric umbilical hernia repair: a prospective randomized clinical trial. JAMA Surg. 2013 Aug;148(8):707-13. doi: 10.1001/jamasurg.2013.1442. PMID 23760519
- [Result] Tomecka MJ, Bortsov AV, Miller NR, Solano N, Narron J, McNaull PP, Ricketts KJ, Lupa CM, McLean SA. Substantial postoperative pain is common among children undergoing laparoscopic appendectomy. Paediatr Anaesth. 2012 Feb;22(2):130-5. doi: 10.1111/j.1460-9592.2011.03711.x. Epub 2011 Sep 29. PMID 21958060
- [Result] Hamill JK, Liley A, Hill AG. Rectus sheath block for laparoscopic appendicectomy: a randomized clinical trial. ANZ J Surg. 2015 Dec;85(12):951-6. doi: 10.1111/ans.12950. Epub 2015 Jan 12. PMID 25581711
- [Result] Hicks CL, von Baeyer CL, Spafford PA, van Korlaar I, Goodenough B. The Faces Pain Scale-Revised: toward a common metric in pediatric pain measurement. Pain. 2001 Aug;93(2):173-183. doi: 10.1016/S0304-3959(01)00314-1. PMID 11427329